CLINICAL TRIAL: NCT02607072
Title: Enteric-coated Aspirin for Prevention of Postsurgical Recurrence and Metastasis in Asian Colorectal Cancer Patients (the APREMEC Trial): a Large-scale Multicenter Randomized Double-blind Placebo-controlled Trial
Brief Title: Aspirin for Prevention of Postsurgical Recurrence and Metastasis in Asian Colorectal Cancer Patients: a Multi-center Randomized Trial
Acronym: APREMEC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Fourth Affiliated Hospital of Anhui Medical University (Other)
Collaborators: The First Affiliated Hospital of Anhui Medical University (Other); Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Lei Huang, Chief doctor, PhD, MD, MSc, MBBS, The Fourth Affiliated Hospital of Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APREMEC-01
Record Dates: First submitted 2015-11-15; First posted 2015-11-17 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Colorectal Cancer
Keywords: APREMEC, aspirin, colorectal cancer, adjuvant therapy, recurrence, metastasis, survival
MeSH Terms: conditions — Colorectal Neoplasms; Recurrence; Neoplasm Metastasis | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Aspirin 200 mg daily (Experimental): Aspirin 200 mg daily
  Interventions: Drug: Acetylsalicylic acid (ASA)/aspirin 200 mg daily
- Aspirin 100 mg daily (Experimental): Aspirin 100 mg daily
  Interventions: Drug: Acetylsalicylic acid (ASA)/aspirin 100 mg daily
- Placebo control (Placebo Comparator): Placebo control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetylsalicylic acid (ASA)/aspirin 200 mg daily
  Arms: Aspirin 200 mg daily
Drug: Acetylsalicylic acid (ASA)/aspirin 100 mg daily
  Arms: Aspirin 100 mg daily
Drug: Placebo
  Arms: Placebo control

SUMMARY:
Background: Evidence of high quality has suggested that acetylsalicylic acid (ASA)/aspirin effectively reduces colorectal adenoma incidence and recurrence rate, and several randomized controlled trials (RCTs) strongly indicate its potential to prevent colorectal cancer (CRC) initiation and progression and to decrease cancer-related mortality. However the role of aspirin supplied as an adjuvant agent in postsurgical CRC patients remains obscure, and a RCT is warranted for clarification.

Aim: The APREMEC trial aims to investigate the potential preventative role of enteric-coated aspirin (100 mg and 200 mg daily) against postsurgical recurrence and metastasis among Asian CRC patients.

Design: The investigators hypothesize that this large-scale multicenter randomized double-blind placebo-controlled trial will support that aspirin can reduce recurrence and metastasis and improve survival in postsurgical non-metastasized CRC patients. The primary endpoint of this trial is disease-free survival, and the secondary endpoints are 3-year and 5-year overall survival, the interactive effects of lifestyle including smoking and alcohol ingestion, and adverse event rate. Eligible postoperative patients with non-metastasized CRC will be randomized in this trial to 100 mg aspirin, 200 mg aspirin or placebo until recurrence/metastasis, severe adverse event, death, or end of study, after standard adjuvant therapy. Individuals with peptic ulcer, bleeding tendency, or previous or ongoing treatment with aspirin or other anticoagulants will be excluded from this trial. Stratification factors are gender, study center, cancer site, and tumor stage. After randomization, patients will be followed up with evaluations at a 3-month interval while taking study drug.

Discussion: This study aims at investigation of aspirin's role as an adjuvant agent in prevention of postsurgical CRC recurrence and metastasis. If results turn out to be positive, Asian and global CRC patients will be greatly benefited, due to the fact that aspirin is inexpensive, easily-accessible, and simply-administered, with well know and managed adverse events.

ELIGIBILITY:
Inclusion Criteria:

* This is a double-blind, placebo-controlled, randomized trial investigating aspirin application in tumor-nodal-metastasis (TNM) stages I-III CRC without metastasis requiring surgical resection. Patients ≥ 18 years who have their primary tumors (and metastatic lymph nodes) completely removed with R0 resection margin, and who have completed standard adjuvant therapy within 3 months without bleeding potential (e.g., platelet count ≥ 100 000/mm3) or other contradictions to aspirin will be eligible for this trial.

Exclusion Criteria:

* Patients allergic to aspirin, receiving previous (within 3 months before surgery) or ongoing treatment with aspirin, other anti-platelet or anticoagulation agent, other Cox inhibitors, glucocorticoid, or drugs severely interfering with aspirin, with peptic ulcer, inflammatory bowel disease (e.g., ulcerative colitis and Crohn's disease), asthma, ischemic heart disease (IHD), class III/IV heart failure (as defined by the New York Heart Association), stroke, thrombotic event, peripheral vascular disease, uncontrolled hypertension, gout or severe liver or renal dysfunction, having undergone coronary artery bypass grafting within 3 months will be excluded from this trial. Other exclusion criteria are: colorectal non-malignant diseases (e.g., familial adenomatous polyposis, and adenoma); recurrent CRC; previous colorectal resection; malignancies other than CRC (excluding non-melanoma skin cancer) within 5 years before intake initiation; pregnancy or nursing; immunosuppressive therapy within 6 months; and enrollment in other CRC clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2015-10; Primary Completion 2020-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China